CLINICAL TRIAL: NCT01256528
Title: A Multidisciplinary Protocol for Planned Skin-Preserving Delayed Breast Reconstruction for Patients With Locally Advanced Breast Cancer Requiring Postmastectomy Radiation Therapy
Brief Title: Delayed-Delayed Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0053; NCI-2011-00270 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Invasive breast carcinoma; Breast reconstruction; Mastectomy; Breast cancer; Delayed-delayed breast reconstruction; Post-mastectomy radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delayed Breast Reconstruction (Experimental): Approximately 3 months after postmastectomy radiation therapy, the preserved, irradiated, and re-inflated breast skin will be used to perform the delayed breast reconstruction. During the stage 2 reconstruction, the implant or expander will be removed and the definitive reconstruction will be performed with the preserved breast skin utilizing a preference for autologous tissue or autologous tissue with an implant due to the potential for complications with implant-based reconstructions after radiation therapy (XRT).
  Interventions: Procedure: Delayed Breast Reconstruction

INTERVENTIONS:
Procedure: Delayed Breast Reconstruction — Approximately 3 months after postmastectomy radiation therapy, the preserved, irradiated, and re-inflated breast skin will be used to perform the delayed breast reconstruction. During the stage 2 reconstruction, the implant or expander will be removed and the definitive reconstruction will be performed with the preserved breast skin utilizing a preference for autologous tissue or autologous tissue with an implant due to the potential for complications with implant-based reconstructions after radiation therapy (XRT).

SUMMARY:
The goal of this clinical research study is to learn if delayed-delayed breast reconstruction in women who require post-mastectomy radiation therapy will improve cosmetic outcomes and result in fewer complications compared to the standard approach (reconstruction that is not started until radiation treatment is completed).

DETAILED DESCRIPTION:
Study Visits and Surgeries:

You will be hospitalized 2-4 times for 1-5 days depending on your condition. If you agree to take part in this study, you will be scheduled for a skin-sparing mastectomy. The following tests and procedures will be performed:

Pre-Operative Visit:

* Your complete medical history will be updated.
* The doctor will determine what type of reconstructive surgery can be done.
* You will have photos taken of your breasts. Your face, hair, or jewelry will not be photographed. These photos will be kept in a password-protected computer accessible only by the principle investigator and people directly involved in this study.
* You will complete a quality of life questionnaire. The questionnaire asks about how satisfied you are with your appearance. The questionnaire will be sent by email, US postal service mail, or in person when you come for your follow up visits. The questionnaire should take about 20 minutes to complete. If sent by US postal service, you will be given a postage-paid envelope to return the questionnaire.

At your Mastectomy Surgery:

* Your complete medical history will be updated.
* You will have photos taken of your breasts.
* During the surgery, a tissue expander will be placed in your breast. Sterile salt water will be added to inflate the expander and a small skin sample (about the size of a pencil eraser) from the breast will be taken to study stretching and scarring of the skin. The tissue will be securely maintained at MD Anderson.
* You will be monitored for any problems.

Post-Operative Visit - 7 to 10 Days after Mastectomy Surgery:

* The study staff will look at the results of your surgery.
* Your complete medical history will be updated.
* You will complete the quality of life questionnaire.
* You will be asked about any problems you may be having.

Deflation Visit - Week 5:

* Your complete medical history will be updated.
* You will have photos taken of your breasts.
* The sterile salt water in the expander will be let out, causing the breast to go flat. This is done by inserting a needle into a special port and withdrawing the fluid with a syringe.

Radiation Visit - Week 8:

* You must have radiation either at M. D. Anderson or an M. D. Anderson-affiliated site.
* Extra fluid may be added to the tissue expander before radiation.
* The study staff will look at the results of your surgery.
* You will be asked about any problems you may be having.
* You will receive radiation, typically 5 days a week for 6 weeks.

Post-Radiation Visits - About Week 13 and every 2 to 4 Weeks after:

* Your complete medical history will be updated.
* The study staff will look at the results of your surgery.
* You will be asked about any problems you may be having.
* You will complete the quality of life questionnaire.
* Your expander will be re-inflated.

Delayed-delayed Reconstruction Surgery - At about Week 23:

* Your complete medical history will be updated.
* You will have photos taken of your breasts.
* During surgery, you will be monitored for any problems. A tissue sample will be collected to study stretching and scarring of the skin from the mastectomy incision and the tissue that is used to form the new breast. The tissue will be securely maintained at MD Anderson.
* During surgery, you will have tissue moved from your lower abdomen, back, or buttock to be used for reconstruction. A silicone or saline breast implant may or may not be used to help construct the breast. The amount of tissue used for building the breast will depend on your body size and donation site. Your reconstructive surgeon will discuss this with you before surgery.
* During surgery, the expander will be removed and reconstruction of your breast will occur.

Follow-Up Surgery - At about Week 47:

* Your complete medical history will be updated.
* You will have photos taken of your breasts.
* You will complete the quality of life questionnaire.
* During surgery, you will be monitored for any problems and a tissue sample will be collected.
* During this surgery, procedures will be done to improve the appearance of the breast.

Long-Term Follow-Up Visits - At 6, 12, 24, and 36 Months:

* Your complete medical history will be updated.
* You will have photos taken of your breasts.
* You will be asked about any problems you may be having.
* At Months 12 and 24, you will complete the quality of life questionnaire.

This is an investigational study. The implants in this study have been FDA approved for skin expansion as a method of breast reconstruction. The use of the implants is investigational in this study.

Up to 200 women will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with invasive breast carcinoma that are scheduled for a mastectomy with planned postmastectomy XRT. This includes, but is not limited to, clinical stage II, III, and IV.
2. Patient must desire breast reconstruction.
3. Patients must sign the informed consent form and must be deemed by operative surgeon not to have medical contraindications for delayed-delayed approach.
4. Patients must be 18 years of age or older.

Exclusion Criteria:

1. Patients in whom it is not known preoperatively to need postmastectomy radiation therapy.
2. Patients with inflammatory breast cancer.
3. Patients in whom the breast skin can not be spared because of involvement with breast cancer.
4. Any patient deemed by the radiation oncologist during preoperative consultation to be an inappropriate patient for this protocol.
5. Patients that can not commit to receiving postmastectomy radiation treatment in addition to breast reconstructive procedures at MD Anderson Cancer Center or satellite affiliates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall Complication Rate | 6 months
  Overall complication defined as any of the following complications post breast reconstruction surgery: seroma, hematoma, wound dehiscence, partial flap loss, total flap loss, infection, flap microvascular thrombosis (arterial or venous), venous congestion of flap, flap fat necrosis, mastectomy skin flap necrosis, exposure breast implant, capsular contracture, and delayed wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Kronowitz, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org